CLINICAL TRIAL: NCT03312270
Title: Strategies to Accommodate Reading (STAR): Using Assistive Technology to Support Reading by People With Aphasia.
Brief Title: Strategies to Accommodate Reading (STAR)
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miami University (Other)
Collaborators: Duquesne University (Other); University of Arizona (Other); Quality Living, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 01446r
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Aphasia
Keywords: aphasia; comprehension; text-to-speech; social validity
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: Examination of comprehension differences when information is presented under different conditions: (a) written only, (b) auditory only or (c) combined written and auditory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodality information Comprehension (Experimental): Evaluate various aspects of multimodality presentation of materials through text-to-speech systems used by people with aphasia.
  Interventions: Behavioral: Multimodality information comprehension

INTERVENTIONS:
Behavioral: Multimodality information comprehension — Evaluate various aspects of multimodality presentation of materials through text-to-speech systems used by people with aphasia.

SUMMARY:
People with aphasia often understand spoken utterances better than written sentences. They also benefit from having content appear in multiple rather than single modalities. Because text-to-speech (TTS) systems accommodate both of these functions, it provides an ideal basis for a reading intervention. TTS systems convert written text to provide both text and auditory information. Research about using TTS supports with people with aphasia has not extended beyond basic case studies and our studies of sentence level comprehension. Hence, no evidence exists about varying TTS features-such as speech output, speech rate, and text highlighting-known to benefit others with reading problems. Also, social acceptance of TTS is not well understood, even though it is critical to adoption and long-term use of the technology.

The purpose of this study is to evaluate various aspects of multimodality presentation of material through TTS systems used by people with aphasia. The immediate outcome of the proposed research will be evidence-based recommendations for selecting and adjusting TTS systems and features. This work will enable clinicians to maximize benefits for adults with varying aphasia profiles. We also will obtain initial evidence about the social validity and perceived value of TTS system use for this population.

DETAILED DESCRIPTION:
Experimental Procedures

* Phase 1: After completing the assessment session, phase one will include up to 4 sessions each lasting up to 90 minutes. Across the four sessions, the participants will listen to and/or read 36 passages ranging from 4 to 6 sentences each. Then, participants will answer 10 multiple choice questions related to the content of the passage. The researcher will provide comprehension support via written choice strategy for the multiple choice questions (e.g., written and spoken language, nonverbal supports such as pointing). Participants will read and/or listen to the stories via a computer. An example of these questions appears in Appendix G.
* Phase 2: After completing the assessment session, phase two will include 1 to 3 separate parts examining 3 different TTS features (e.g., speech presentation rate, text highlighting, speech production quality). Participants can choose to participate in 1 or more parts within this phase. For each part, participants will first listen to or view selected variations of a target feature and choose their preferred variation. For each study, participants will then complete five or four experimental sessions lasting up to 90 minutes each. Parts with up to five sessions (i.e., Part 1 and 2) will include features with more variations than those included in Part 3, which will include up to four sessions. Participants will read and/or listen to up to 12 reading passages in each session and answer multiple choice comprehension questions related to the content of the passage. At the conclusion of each session, participants will provide their opinion about the optimal targeted feature variation using rating forms and interview questions. Participants will read and/or listen to the passages via a computer.
* Phase 3: After completing the assessment session and any previous study phases, the participants will complete one 2-hour session. Participants will complete three activities: (1) education and system exploration guided by a member of the research team, (2) satisfaction and predicted use ratings of TTS systems, and (3) semi-structured interviews. Ratings of the TTS systems will be complete using Likert ratings scales (see Appendix H). Semi-structured interview questions will relate to rationales for system ratings and perceived application of TTS systems for functional use.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of aphasia with reading comprehension impairment resulting from stroke
* Age 19-90 years
* At least 6 months post stroke
* American English is primary language

Exclusion Criteria:

* Presence of hearing impairment (i.e., prescribed bilateral hearing aids or failed hearing screening)
* Presence of vision or motor impairments as determined by screening task described below.
* History of neurological or developmental (reading or learning) impairment other than stroke as determined by self- or family-report.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
1. What is the accuracy with which people with aphasia comprehend paragraph-level information presented as single modalities (auditory or written) versus multiple modalities (written and auditory)? | 4 sessions, 9 minutes each over the course of 1 month
  Participants will answer questions after listening and/or reading stories

SECONDARY OUTCOMES:
Which text-to-speech systems feature variations do people with aphasia prefer and derive the most benefit in terms of comprehension accuracy? | Up to 5 sessions, 90 minutes each over the course of 1 month
  Read stories, answer multiple choice questions. Identify feature preferences.
3. How do people with aphasia perceive and behave when using currently available text-to-speech systems? | 1 session lasting up to 2 hours
  Participants will learn about text-to-speech systems and complete interview about preferences

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Knollman-Porter, PhD, Principal Investigator — Miami University
Locations (2):
- United States (2):
  - Miami University, Oxford, Ohio
  - Duquesne University, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
We will not be sharing the data because of possible breach of privacy given the small number of local people with aphasia.